CLINICAL TRIAL: NCT02057211
Title: Mesenchymal Stem Cells to Intervene in the Development of Type 1 Diabetes: a Blinded Randomized Study
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Changed regulations of culture procedure
Sponsor: Uppsala University Hospital (Other)
Responsible Party: Principal Investigator, Per-Ola Carlsson, Professor, Uppsala University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: AS Dnr2013/195
Record Dates: First submitted 2014-02-04; First posted 2014-02-07 (Estimated); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- sham transplantation of mesenchymal stem cells (Placebo Comparator): control arm with sham transplantation
  Interventions: Procedure: sham transplantation of mesenchymal stem cells
- autologous mesenchymal stem cell transplantation (Active Comparator): Active arm with transplantation of cells
  Interventions: Biological: autologous mesenchymal stem cell transplantation

INTERVENTIONS:
Biological: autologous mesenchymal stem cell transplantation
  Arms: autologous mesenchymal stem cell transplantation
Procedure: sham transplantation of mesenchymal stem cells — Placebo control for transplantation of mesenchymal stem cells
  Arms: sham transplantation of mesenchymal stem cells

SUMMARY:
This project aims to evaluate the efficacy of autologous mesenchymal stem cell treatment to preserve insulin production and beta-cell mass in recently diagnosed patients with type 1 diabetes mellitus. The hypothesis to be tested is that an increased number of circulating mesenchymal stem cells will provide immune modulatory properties, and thereby stop the immune process in islets causing progressive beta-cell death.

ELIGIBILITY:
Inclusion Criteria:

* fasting C-peptide >0.12 nmol/l
* within three weeks of diagnosis of type 1 diabetes

Exclusion Criteria:

* body mass index (BMI) >30
* unstable cardiovascular status incl. New York Heart Association (NYHA) class III/IV
* patients with known or previous malignancy
* active infections incl. serological evidence of infection with HIV, Treponema pallidum, hepatitis B (patients with serology consistent with previous vaccination and a history of vaccination are acceptable) or hepatitis C.
* immune suppressive treatment
* women being pregnant or nursing, or women physiologically capable of becoming pregnant, unless they are using effective methods of contraception during study

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
∆-change of C-peptide Area Under the Curve (AUC) (0-120 min) for a mixed meal tolerance test at two year follow-up when compared to pre-treatment values at enrolment. | ∆-change will be assessed as a difference between two years after transplantation/sham transplantation of mesenchymal stem cells when compared to before transplantation/sham transplantation, i.e. at time 0.

CONTACTS AND LOCATIONS:
Overall Officials: Per-Ola Carlsson, MD, PhD, Principal Investigator — Uppsala University Hospital
Locations (1):
- Uppsala University Hospital, Uppsala, Sweden